CLINICAL TRIAL: NCT00432276
Title: A Multicenter, Randomized, Double-Blind Study to Determine the Efficacy and Safety of the Addition of SYR-322 25 mg Versus Dose Titration From 30 mg to 45 mg of Pioglitazone HCl (ACTOS®) in Subjects With Type 2 Diabetes Mellitus Who Have Inadequate Control on a Combination of Metformin and 30 mg of Pioglitazone HCl Therapy
Brief Title: Efficacy of Alogliptin and Pioglitazone in Subjects With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 01-06-TL-322OPI-004; 2006-006025-73 (EudraCT Number); U1111-1112-3363 (Other: WHO)
Record Dates: First submitted 2007-02-05; First posted 2007-02-07 (Estimated); Results first posted 2013-04-04 (Estimated); Last update posted 2013-04-04 (Estimated); Status verified 2013-04

CONDITIONS: Diabetes Mellitus
Keywords: Glucose Metabolism Disorder; Dysmetabolic Syndrome; Type II Diabetes; Diabetes Mellitus, Lipoatrophic; Dyslipidemia; Hyperglycemia; Drug Therapy
MeSH Terms: conditions — Diabetes Mellitus; Glucose Metabolism Disorders; Diabetes Mellitus, Type 2; Diabetes Mellitus, Lipoatrophic; Dyslipidemias; Hyperglycemia | interventions — alogliptin; Pioglitazone; Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Alogliptin 25 mg + Pioglitazone 30 mg add-on to Metformin (Experimental): Alogliptin 25 mg, tablets, orally, once daily; pioglitazone 30 mg, tablets, orally, once daily; and the maximum tolerated dose of metformin, tablets, orally, for up to 52 weeks.
  Interventions: Drug: Alogliptin; Drug: Pioglitazone; Drug: Metformin; Drug: Placebo
- Pioglitazone 45 mg add-on to Metformin (Active Comparator): Alogliptin placebo-matching tablets, orally, once daily; pioglitazone 45 mg, tablets, orally, once daily; and the maximum tolerated dose of metformin, tablets, orally, for up to 52 weeks.
  Interventions: Drug: Pioglitazone; Drug: Metformin; Drug: Placebo

INTERVENTIONS:
Drug: Alogliptin — Alogliptin tablets.
  Other Names: SYR-322
  Arms: Alogliptin 25 mg + Pioglitazone 30 mg add-on to Metformin
Drug: Pioglitazone — Pioglitazone tablets.
  Other Names: ACTOS®
Drug: Metformin — Metformin HCl tablets (immediate-release, commercially available formulation) ≥1500 mg or maximum tolerated dose.
Drug: Placebo — Matching placebo tablets.

SUMMARY:
The purpose of the study is to compare the effect of adding alogliptin, once daily (QD), to the ongoing treatment regimen of pioglitazone HCl and metformin in patients with inadequate glycemic control.

DETAILED DESCRIPTION:
Despite the introduction of new classes of medications for glycemic control, just over half of adults with type 2 diabetes mellitus (T2DM) achieve a glycosylated hemoglobin level less than 7.0%, the American Diabetes Association recommended glycosylated hemoglobin goal. The rising incidence of type 2 diabetes mellitus along with limitations of the currently available treatments suggest the need for new therapies for glycemic control along with the increased requirement for combination therapy in type 2 diabetes mellitus.

Thiazolidinediones increase glucose utilization, decrease gluconeogenesis, and increase glucose disposal through an incompletely understood mechanism but one associated with binding of the drug to nuclear receptors known as peroxisome proliferator-activated receptors-gamma. Peroxisome proliferator-activated receptors-gamma are found in tissues important for insulin action, such as adipose tissue, skeletal muscle, and the liver. The greatest concentration of peroxisome proliferator-activated receptors-gamma receptors is in adipose tissue. Thiazolidinediones reduce insulin resistance by enhancing insulin sensitivity in muscle cells, adipose tissue, and hepatic cells (inhibiting hepatic gluconeogenesis) with no direct impact on insulin secretion. Thus, thiazolidinediones improve glycemic control and result in reduced levels of circulating insulin. Pioglitazone HCl (ACTOS®) is a thiazolidinedione developed by Takeda Chemical Industries, Ltd. (Osaka, Japan). Pioglitazone depends on the presence of insulin for its mechanism of action. Worldwide clinical investigation has shown that, as an adjunct to diet and exercise, pioglitazone improves glycemic control when used as monotherapy, and in combination with commonly used antidiabetic medications (ie, sulfonylureas, metformin, or insulin).

SYR-322 (alogliptin) is a selective, orally available inhibitor of dipeptidyl peptidase IV currently in development by Takeda Global Research & Development Center, Inc. as a treatment for type 2 diabetes mellitus. Dipeptidyl peptidase IV is the primary enzyme involved in the in vivo degradation of at least 2 peptide hormones released in response to nutrient ingestion, namely glucagon-like peptide-1 and glucose-dependent insulinotropic peptide. Both peptides exert important effects on islet β-cells to stimulate glucose-dependent insulin secretion and regulate β-cell proliferation and cytoprotection. Glucagon-like peptide-1 also inhibits gastric emptying, glucagon secretion, and food intake. The glucose-lowering actions of glucagon-like peptide-1, but not glucose-dependent insulinotropic peptide, are preserved in patients with type 2 diabetes.

Given the complementary mechanisms of action of alogliptin (stimulation of insulin secretion) and pioglitazone (enhancement of insulin sensitivity) and the absence of overlapping safety risks, the introduction of this combination therapy in patients with T2DM could potentially show enhanced glycemic control and allow patients to reach and maintain their HbA1c goal more effectively.

This study is designed to determine if the addition of alogliptin to a combination of pioglitazone with metformin can be effective at achieving glycemic control without increasing safety risks versus the titration of pioglitazone to 45 mg with metformin in patients with type 2 diabetes mellitus who are experiencing inadequate glycemic control on a current regimen of metformin.

ELIGIBILITY:
Inclusion Criteria:

* Has a historical diagnosis of type 2 diabetes mellitus.
* Meets one of the following:

  * Has been inadequately controlled (HbA1c between 7% and 10%, inclusive) on a stable dose of greater than or equal to 1500 mg (or maximum tolerated dose) of metformin and 30 mg of pioglitazone
  * Has been inadequately controlled (as defined by an HbA1c ≥7.5%) on a combination therapy including metformin and another oral antidiabetic agent (ie, sulfonylureas, rosiglitazone maleate, or pioglitazone 15 mg, etc). Subjects on a combination therapy that included a DPP-4 inhibitor were excluded.
* No treatment with antidiabetic agents other than metformin and pioglitazone.
* Body mass index greater than or equal to 23 kg/m^2 and less than or equal to 45 kg/m^2.
* Fasting plasma C-peptide concentration greater than or equal to 0.8 ng/mL.
* Systolic blood pressure less than 160 mmHg and diastolic pressure less than 100 mmHg.
* Hemoglobin greater than or equal to 12 g/dL for males and greater than or equal to 10 g/dL for females.
* Alanine aminotransferase less than or equal to 2.5 x upper limit of normal.
* Serum creatinine less than 1.5 mg/dL for males and less than 1.4 mg/dL for females.
* Thyroid-stimulating hormone level less than or equal to the upper limit of normal range and the patient is clinically euthyroid.
* Females of childbearing potential who are sexually active must agree to use adequate contraception, and can neither be pregnant nor lactating from Screening throughout the duration of the study.
* Able and willing to monitor their own blood glucose concentrations with a home glucose monitor.
* No major illness or debility that in the investigator's opinion prohibits the patient from completing the study.

Exclusion Criteria:

* Urine albumin/creatinine ratio of greater than 1000 μg/mg.
* History of cancer, other than squamous cell or basal cell carcinoma of the skin, that has not been in full remission for at least 5 years prior to Screening.
* History of bladder cancer.
* History of laser treatment for proliferative diabetic retinopathy within the 6 months prior to Screening.
* Patients with unexplained microscopic hematuria of greater than +1, confirmed by repeat testing.
* History of treated diabetic gastroparesis.
* History of gastric bypass surgery.
* New York Heart Association Class I-IV heart failure regardless of therapy.
* History of coronary angioplasty, coronary stent placement, coronary bypass surgery, or myocardial infarction within the 6 months prior to Screening.
* History of any hemoglobinopathy that may affect determination of glycosylated hemoglobin.
* History of infection with hepatitis B, hepatitis C, or human immunodeficiency virus.
* History of a psychiatric disorder that will affect the patient's ability to participate in the study.
* History of angioedema in association with use of angiotensin-converting enzyme inhibitors or angiotensin-II receptor inhibitors.
* History of alcohol abuse or substance abuse within the 2 years prior to Screening.
* Receipt of any investigational drug within the 30 days prior to Screening or a history of receipt of an investigational antidiabetic drug within the 3 months prior to Screening.
* Prior treatment in an investigational study of alogliptin.
* Hypersensitive to pioglitazone HCl, metformin, alogliptin or other excipients.
* The patient has donated more than 400 mL of blood within the 90 days prior to Screening and Pre-Screening, if applicable.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 803 (Actual)
Dates: Start 2007-01; Primary Completion 2009-05 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: VP Biological Sciences, Study Director — Takeda
Locations (86):
- United States (86):
  - Birmingham, Alabama
  - Huntsville, Alabama
  - Lake Havasu City, Arizona
  - Little Rock, Arkansas
  - Foothill Ranch, California
  - Los Alamitos, California
  - Los Angeles, California
  - Pismo Beach, California
  - San Diego, California
  - Golden, Colorado
  - Clearwater, Florida
  - Hialeah, Florida
  - Lakeland, Florida
  - Marianna, Florida
  - Miami, Florida
  - North Miami Beach, Florida
  - Pembroke Pines, Florida
  - Sebastian, Florida
  - South Miami, Florida
  - Tampa, Florida
  - Winter Park, Florida
  - Blue Ridge, Georgia
  - Conyers, Georgia
  - Decatur, Georgia
  - Duluth, Georgia
  - Dunwoody, Georgia
  - Warner Robins, Georgia
  - Boise, Idaho
  - Coeur d'Alene, Idaho
  - Burr Ridge, Illinois
  - Chicago, Illinois
  - Melrose Park, Illinois
  - Naperville, Illinois
  - O'Fallon, Illinois
  - Bloomington, Indiana
  - Mishawaka, Indiana
  - Overland Park, Kansas
  - Marrero, Louisiana
  - Elkton, Maryland
  - Rockville, Maryland
  - Towson, Maryland
  - Marlborough, Massachusetts
  - Bay City, Michigan
  - Saint Clair Shores, Michigan
  - McCook, Nebraska
  - Las Vegas, Nevada
  - Blackwood, New Jersey
  - Trenton, New Jersey
  - West Caldwell, New Jersey
  - Asheboro, North Carolina
  - Charlotte, North Carolina
  - Mooresville, North Carolina
  - Shelby, North Carolina
  - Sparta, North Carolina
  - Bismarck, North Dakota
  - Orrville, Ohio
  - Norman, Oklahoma
  - Ashland, Oregon
  - Aliquippa, Pennsylvania
  - Altoona, Pennsylvania
  - Dawningtown, Pennsylvania
  - Fleetwood, Pennsylvania
  - Kingston, Pennsylvania
  - Norristown, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Tipton, Pennsylvania
  - Florence, South Carolina
  - Taylors, South Carolina
  - Williamston, South Carolina
  - Watertown, South Dakota
  - Kingsport, Tennessee
  - Milan, Tennessee
  - Nashville, Tennessee
  - Arlington, Texas
  - Austin, Texas
  - Colleyville, Texas
  - El Paso, Texas
  - Garland, Texas
  - Houston, Texas
  - Hurst, Texas
  - San Antonio, Texas
  - Seguin, Texas
  - Hampton, Virginia
  - Norfolk, Virginia
  - Richmond, Virginia
  - Virginia Beach, Virginia

REFERENCES:
- [Result] Bosi E, Ellis GC, Wilson CA, Fleck PR. Alogliptin as a third oral antidiabetic drug in patients with type 2 diabetes and inadequate glycaemic control on metformin and pioglitazone: a 52-week, randomized, double-blind, active-controlled, parallel-group study. Diabetes Obes Metab. 2011 Dec;13(12):1088-96. doi: 10.1111/j.1463-1326.2011.01463.x. PMID 21733058
- See also: ACTOS® Package Insert — http://general.takedapharm.com/content/file/pi.pdf?applicationcode=ab2d7112-8eb3-465a-8fda-35018a9eafb0&fileTypeCode=ACTOSPI

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 235 investigative sites in 16 countries worldwide from 30 January 2007 to 5 June 2009.
Pre-assignment Details: Participants with a diagnosis of type 2 diabetes who were experiencing inadequate glycemic control on their existing treatment regimen of metformin HCl plus pioglitazone were randomized in a 1:1 ratio to 1 of 2 treatment arms: addition of alogliptin 25 mg versus titration of pioglitazone 30 mg to 45 mg.
Groups:
- Alogliptin 25 mg + Pioglitazone 30 mg + Metformin: Alogliptin 25 mg, tablets, orally, once daily; pioglitazone 30 mg, tablets, orally, once daily; and the maximum tolerated dose of metformin, tablets, orally, for up to 52 weeks.
- Pioglitazone 45 mg + Metformin: Alogliptin placebo-matching tablets, orally, once daily; pioglitazone 45 mg, tablets, orally, once daily; and the maximum tolerated dose of metformin, tablets, orally, for up to 52 weeks.
Period: Overall Study
Arm/Group | Alogliptin 25 mg + Pioglitazone 30 mg + Metformin | Pioglitazone 45 mg + Metformin
Started | 404 | 399
Per Protocol Set | 303 (Patients who received at least 1 dose of study medication and who had no major protocol violations.) | 306
Completed | 283 | 243
Not Completed | 121 | 156
Not completed — Hyperglycemic Rescue | 44 | 87
Not completed — Adverse Event | 13 | 16
Not completed — Protocol Violation | 25 | 20
Not completed — Lost to Follow-up | 6 | 2
Not completed — Withdrawal by Subject | 25 | 20
Not completed — Physician Decision | 6 | 8
Not completed — Other | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Alogliptin 25 mg + Pioglitazone 30 mg + Metformin | Pioglitazone 45 mg + Metformin | Total
Number analyzed (Participants) | 404 | 399 | 803
Age Continuous [Mean (Standard Deviation); unit: years] | 54.3 (9.86) | 55.9 (9.94) | 55.1 (9.93)
Age, Customized [Number; unit: participants]
  <65 years | 339 | 320 | 659
  ≥65 years | 65 | 79 | 144
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 194 | 195 | 389
  Male | 210 | 204 | 414
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 30 | 31 | 61
  Not Hispanic or Latino | 374 | 368 | 742
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian or Alaska Native | 2 | 0 | 2
  Asian | 79 | 78 | 157
  Black or African American | 41 | 36 | 77
  Native Hawaiian or Other Pacific Islander | 2 | 0 | 2
  White | 242 | 256 | 498
  Other | 38 | 29 | 67
Height [Mean (Standard Deviation); unit: cm] | 166.82 (9.884) | 166.37 (10.856) | 166.60 (10.375)
Weight [Mean (Standard Deviation); unit: kg] | 88.16 (18.898) | 87.98 (19.283) | 88.07 (19.078)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 31.52 (5.248) | 31.58 (5.177) | 31.55 (5.210)
Duration of diabetes [Mean (Standard Deviation); unit: years] | 7.47 (5.243) | 6.85 (4.611) | 7.16 (4.946)
Baseline daily metformin HCl use [Median (Full Range); unit: mg] | 1700.0 [500 to 3400] | 1700.0 [500 to 3000] | 1700.0 [500 to 3400]
Current smoker [Number; unit: participants]
  Yes | 100 | 99 | 199
  No | 304 | 300 | 604
HbA1c [Number; unit: participants] — HbA1c category is based on HbA1c value used in randomization for stratification.
  participants
    <8.0% | 161 | 163 | 324
    ≥8.0% | 243 | 236 | 479

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Glycosylated Hemoglobin (HbA1c)
Description: The change from Baseline to Week 26 and Week 52 in HbA1c (the concentration of glucose bound to hemoglobin as a percent of the absolute maximum that can be bound).
Time Frame: Baseline and Weeks 26 and 52.
Population: Per-protocol set included all randomized patients who received at least 1 dose of double-blind study medication and who had no major protocol violations. Last observation carried forward (LOCF) imputation was utilized.
Measure: Least Squares Mean (Standard Error); unit: percentage of glycosylated hemoglobin
Arm/Group | Alogliptin 25 mg + Pioglitazone 30 mg + Metformin | Pioglitazone 45 mg + Metformin
Number analyzed (Participants) | 303 | 306
percentage of glycosylated hemoglobin
  Change from Baseline at Week 26 | -0.89 (0.042) | -0.42 (0.042)
  Change from Baseline at Week 52 | -0.70 (0.048) | -0.29 (0.048)
Statistical Analysis 1: Comparison: Alogliptin 25 mg + Pioglitazone 30 mg + Metformin vs Pioglitazone 45 mg + Metformin; The analysis was conducted at the 1-sided 0.025 significance level. Non-inferiority was demonstrated if the upper confidence limit for the LS mean difference was less than +0.3%; Test type: Non-Inferiority or Equivalence — The analysis was conducted at the 1-sided 0.025 significance level. Non-inferiority was demonstrated if the upper confidence limit for the LS mean difference was less than +0.3%; ANCOVA; LS mean difference = -0.47, 97.5% CI 1-sided [upper limit -0.35] — Least squares means are from an ANCOVA model with treatment, study schedule, and geographic region as class variables, and baseline metformin dose and baseline HbA1c as covariates
Statistical Analysis 2: Comparison: Alogliptin 25 mg + Pioglitazone 30 mg + Metformin vs Pioglitazone 45 mg + Metformin; Comparison of Change from Baseline at Week 52. The null hypothesis was that the average change from Baseline in HbA1c at Week 52 for the alogliptin 25 mg addition group is inferior to the average change for the pioglitazone titration group. The alternative hypothesis was that the change from Baseline in HbA1c for the alogliptin 25 mg addition group was non-inferior to the change for the pioglitazone titration group for at Week 52; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ANCOVA; LS mean difference = -0.42, 97.5% CI 1-sided [upper limit -0.28] — [estimate comment as in outcome 1, analysis 1]

2. Secondary Outcome: Change From Baseline in HbA1c Over Time
Description: The change from Baseline in HbA1c (the concentration of glucose bound to hemoglobin as a percent of the absolute maximum that can be bound) during the study. Least Squares Means were from an Analysis of Covariance (ANCOVA) model with treatment, study schedule, and geographic region as class variables, and baseline metformin dose and baseline HbA1c as covariates.
Time Frame: Baseline and Weeks 4, 8, 12, 16, 20, 34 and 42.
Population: Per-protocol set. Last observation carried forward (LOCF) imputation was utilized.
Measure: Least Squares Mean (Standard Error); unit: percentage of glycosylated hemoglobin
Arm/Group | Alogliptin 25 mg + Pioglitazone 30 mg + Metformin | Pioglitazone 45 mg + Metformin
Number analyzed (Participants) | 303 | 306
percentage of glycosylated hemoglobin
  Change from Baseline at Week 4 (n=276, 277) | -0.42 (0.025) | -0.15 (0.025)
  Change from Baseline at Week 8 (n=303, 306) | -0.71 (0.030) | -0.27 (0.030)
  Change from Baseline at Week 12 (n=303, 306) | -0.85 (0.037) | -0.35 (0.037)
  Change from Baseline at Week 16 (n=303, 306) | -0.91 (0.039) | -0.43 (0.038)
  Change from Baseline at Week 20 (n=303, 306) | -0.91 (0.039) | -0.45 (0.039)
  Change from Baseline at Week 34 (n=303, 306) | -0.82 (0.046) | -0.37 (0.045)
  Change from Baseline at Week 42 (n=303, 306) | -0.80 (0.048) | -0.36 (0.048)
Statistical Analysis 1: Comparison: Alogliptin 25 mg + Pioglitazone 30 mg + Metformin vs Pioglitazone 45 mg + Metformin; Comparison of change from Baseline in HbA1c at Week 42; Test type: Superiority or Other; p < 0.001, ANCOVA — Statistical tests and resulting P-values are 2-sided and was evaluated at the 0.05 significance level; ANCOVA model with treatment, study schedule, and geographic region as class variables, and baseline metformin dose and baseline HbA1c as covariates; LS Mean Difference = -0.44, 95% CI 2-sided [-0.57 to -0.31]

3. Secondary Outcome: Percentage of Participants With Glycosylated Hemoglobin ≤ 6.5%
Description: Clinical response at Weeks 26 and 52 was assessed by the percentage of participants with HbA1c less than or equal to 6.5%.
Time Frame: Weeks 26 and 52.
Population: The full analysis set. Patients who did not complete the scheduled Week 26 or Week 52 visit were assessed based on their response at the time of discontinuation.
Measure: Number; unit: percentage of participants
Arm/Group | Alogliptin 25 mg + Pioglitazone 30 mg + Metformin | Pioglitazone 45 mg + Metformin
Number analyzed (Participants) | 404 | 399
percentage of participants
  Week 26 | 13.9 | 7.8
  Week 52 | 8.7 | 4.3

4. Secondary Outcome: Percentage of Participants With Glycosylated Hemoglobin ≤ 7.0%
Description: Clinical response at Weeks 26 and 52 was assessed by the percentage of participants with HbA1c less than or equal to 7%.
Time Frame: Weeks 26 and 52.
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Alogliptin 25 mg + Pioglitazone 30 mg + Metformin | Pioglitazone 45 mg + Metformin
Number analyzed (Participants) | 404 | 399
percentage of participants
  Week 26 | 39.1 | 25.8
  Week 52 | 33.2 | 21.3

5. Secondary Outcome: Percentage of Participants With Glycosylated Hemoglobin ≤ 7.5%
Description: Clinical response at Weeks 26 and 52 was assessed by the percentage of participants with HbA1c less than or equal to 7.5%.
Time Frame: Weeks 26 and 52.
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Alogliptin 25 mg + Pioglitazone 30 mg + Metformin | Pioglitazone 45 mg + Metformin
Number analyzed (Participants) | 404 | 399
percentage of participants
  Week 26 | 64.9 | 47.1
  Week 52 | 59.9 | 44.1

6. Secondary Outcome: Percentage of Participants With a Decrease in Glycosylated Hemoglobin ≥ 0.5%
Description: Clinical response at Weeks 26 and 52 was assessed by the percentage of participants with a decrease from Baseline in HbA1c of greater than or equal to 0.5%.
Time Frame: Weeks 26 and 52.
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Alogliptin 25 mg + Pioglitazone 30 mg + Metformin | Pioglitazone 45 mg + Metformin
Number analyzed (Participants) | 404 | 399
percentage of participants
  Week 26 | 72.0 | 42.1
  Week 52 | 60.9 | 37.6

7. Secondary Outcome: Percentage of Participants With a Decrease in Glycosylated Hemoglobin ≥ 1.0%
Description: Clinical response at Weeks 26 and 52 was assessed by the percentage of participants with a decrease from Baseline in HbA1c of greater than or equal to 1.0%.
Time Frame: Weeks 26 and 52.
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Alogliptin 25 mg + Pioglitazone 30 mg + Metformin | Pioglitazone 45 mg + Metformin
Number analyzed (Participants) | 404 | 399
percentage of participants
  Week 26 | 42.3 | 20.3
  Week 52 | 35.6 | 17.3

8. Secondary Outcome: Percentage of Participants With a Decrease in Glycosylated Hemoglobin ≥ 1.5%
Description: Clinical response at Weeks 26 and 52 was assessed by the percentage of participants with a decrease from Baseline in HbA1c of greater than or equal to 1.5%.
Time Frame: Weeks 26 and 52.
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Alogliptin 25 mg + Pioglitazone 30 mg + Metformin | Pioglitazone 45 mg + Metformin
Number analyzed (Participants) | 404 | 399
percentage of participants
  Week 26 | 18.6 | 7.5
  Week 52 | 17.1 | 8.0

9. Secondary Outcome: Percentage of Participants With a Decrease in Glycosylated Hemoglobin ≥ 2.0%
Description: Clinical response at Weeks 26 and 52 was assessed by the percentage of participants with a decrease from Baseline in HbA1c of greater than or equal to 2.0%.
Time Frame: Weeks 26 and 52.
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Alogliptin 25 mg + Pioglitazone 30 mg + Metformin | Pioglitazone 45 mg + Metformin
Number analyzed (Participants) | 404 | 399
percentage of participants
  Week 26 | 8.2 | 3.0
  Week 52 | 7.9 | 3.3

10. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose
Description: The change from Baseline in fasting plasma glucose (FPG) was assessed at Weeks 2, 4, 8, 12, 16, 20, 26, 34, 42 and 52. Least Squares Means were from an ANCOVA model with treatment, study schedule and geographic region as class variables, and baseline metformin dose and baseline FPG as covariates.
Time Frame: Baseline and Weeks 2, 4, 8, 12, 16, 20, 26, 34, 42 and 52.
Population: The full analysis set, which included all randomized patients who received at least 1 dose of double-blind study drug and where Baseline and at least 1 postbaseline value were available. Last observation carried forward (LOCF) imputation was utilized.
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Alogliptin 25 mg + Pioglitazone 30 mg + Metformin | Pioglitazone 45 mg + Metformin
Number analyzed (Participants) | 404 | 399
mg/dL
  Week 2 (n=360, 345) | -15.5 (1.56) | -0.5 (1.59)
  Week 4 (n=397, 394) | -17.7 (1.48) | -1.4 (1.49)
  Week 8 (n=399, 396) | -19.1 (1.56) | -5.7 (1.57)
  Week 12 (n=399, 396) | -19.6 (1.60) | -4.8 (1.61)
  Week 16 (n=399, 396) | -18.0 (1.60) | -4.5 (1.60)
  Week 20 (n=399, 396) | -16.4 (1.65) | -5.8 (1.66)
  Week 26 (n=399, 396) | -17.1 (1.79) | -4.9 (1.79)
  Week 34 (n=399, 396) | -13.6 (1.88) | -6.2 (1.88)
  Week 42 (n=399, 396) | -15.9 (1.87) | -4.9 (1.88)
  Week 52 (n=399, 396) | -14.6 (1.89) | -3.7 (1.89)
Statistical Analysis 1: Comparison: Alogliptin 25 mg + Pioglitazone 30 mg + Metformin vs Pioglitazone 45 mg + Metformin; Comparison of change from Baseline at Week 52; Test type: Superiority or Other; p < 0.001, ANCOVA — Statistical test and resulting P-value are 2-sided and was evaluated at the 0.05 significance level; ANCOVA model with treatment, study schedule and geographic region as class variables, and baseline metformin dose and FPG as covariates; LS Mean Difference = -10.9, 95% CI 2-sided [-16.2 to -5.7]

11. Secondary Outcome: Percentage of Participants With Marked Hyperglycemia
Description: Marked Hyperglycemia is defined as fasting plasma glucose greater than or equal to 200 mg/dL (11.10 mmol/L).
Time Frame: Baseline to Week 52
Population: Full Analysis Set including patients with at least one non-missing fasting plasma glucose result in each treatment group.
Measure: Number; unit: percentage of participants
Arm/Group | Alogliptin 25 mg + Pioglitazone 30 mg + Metformin | Pioglitazone 45 mg + Metformin
Number analyzed (Participants) | 399 | 396
percentage of participants | 27.3 | 36.1
Statistical Analysis 1: Comparison: Alogliptin 25 mg + Pioglitazone 30 mg + Metformin vs Pioglitazone 45 mg + Metformin; Comparison of incidence of marked hyperglycemia through Week 52; Test type: Superiority or Other; p < 0.001, Extended Mantel Haenszel Test — Statistical test and resulting P-value are 2-sided and was evaluated at the 0.05 significance level; Treatment comparison was performed using nonparametric, covariance-adjusted, extended Mantel-Haenszel test

12. Secondary Outcome: Percentage of Participants Meeting Hyperglycemic Rescue Criteria
Description: Rescue was defined as meeting 1 of the following criteria, confirmed by a 2nd sample drawn within 7 days after the first sample and analyzed by the central laboratory:
  1. After more than 2 weeks of treatment but prior to the Week 4 Visit: A single fasting plasma glucose (FPG) ≥275 mg/dL;
  2. From the Week 4 Visit but prior to the Week 8 Visit: A single FPG ≥250 mg/dL;
  3. From the Week 8 Visit but prior to the Week 12 Visit: A single FPG ≥225 mg/dL;
  4. From the Week 12 Visit through the End-of-Treatment Visit: HbA1c ≥8.5% AND ≤0.5% reduction in HbA1c as compared with the baseline HbA1c.
Time Frame: Baseline to Week 52
Population: Full Analysis Set including patients with a postbaseline visit.
Measure: Number; unit: percentage of participants
Arm/Group | Alogliptin 25 mg + Pioglitazone 30 mg + Metformin | Pioglitazone 45 mg + Metformin
Number analyzed (Participants) | 402 | 397
percentage of participants | 10.9 | 21.7
Statistical Analysis 1: Comparison: Alogliptin 25 mg + Pioglitazone 30 mg + Metformin vs Pioglitazone 45 mg + Metformin; Comparison of incidence of hyperglycemic rescue through Week 52; Test type: Superiority or Other; p < 0.001, Extended Mantel Haenszel Test — Statistical test and resulting P-value are 2-sided and was evaluated at the 0.05 significance level; Treatment comparison was performed using nonparametric, covariance-adjusted, extended Mantel-Haenszel test

13. Secondary Outcome: Change From Baseline in Fasting Proinsulin
Description: Proinsulin is a precursor to insulin, and was measured as an indicator of pancreatic function. The change from Baseline in fasting proinsulin was assessed at Weeks 4, 8, 12, 16, 20, 26, 34, 42 and 52. Least Squares Means were from an ANCOVA model with treatment, study schedule and geographic region as class variables, and baseline metformin dose and baseline fasting proinsulin as covariates.
Time Frame: Baseline and Weeks 4, 8, 12, 16, 20, 26, 34, 42 and 52.
Population: The full analysis set where Baseline and at least 1 postbaseline value were available. Last observation carried forward (LOCF) imputation was utilized.
Measure: Least Squares Mean (Standard Error); unit: pmol/L
Arm/Group | Alogliptin 25 mg + Pioglitazone 30 mg + Metformin | Pioglitazone 45 mg + Metformin
Number analyzed (Participants) | 404 | 399
pmol/L
  Week 4 (n=342, 325) | -2.0 (0.67) | -0.8 (0.69)
  Week 8 (n=380, 376) | -2.3 (0.77) | -0.5 (0.77)
  Week 12 (n=380, 376) | -1.3 (0.89) | 1.6 (0.89)
  Week 16 (n=381, 376) | -0.2 (1.01) | 0.6 (1.02)
  Week 20 (n=381, 376) | -0.5 (0.67) | 0.3 (0.68)
  Week 26 (n=381, 376) | 0.6 (0.82) | 0.7 (0.83)
  Week 34 (n=381, 376) | 0.9 (0.86) | 0.3 (0.86)
  Week 42 (n=381, 376) | -0.1 (0.80) | 1.1 (0.81)
  Week 52 (n=381, 376) | -0.5 (0.74) | 1.2 (0.74)
Statistical Analysis 1: Comparison: Alogliptin 25 mg + Pioglitazone 30 mg + Metformin vs Pioglitazone 45 mg + Metformin; Comparison of change from Baseline at Week 52; Test type: Superiority or Other; p = 0.116, ANCOVA — Statistical test and resulting P-value are 2-sided and was evaluated at the 0.05 significance level; ANCOVA model with treatment, study schedule and geographic region as class variables, and baseline metformin dose and proinsulin as covariates; LS Mean Difference = -1.6, 95% CI 2-sided [-3.7 to 0.4]

14. Secondary Outcome: Change From Baseline in Fasting Insulin
Description: The change from Baseline in fasting insulin was assessed at Weeks 4, 8, 12, 16, 20, 26, 34, 42 and 52. Least Squares Means were from an ANCOVA model with treatment, study schedule and geographic region as class variables, and baseline metformin dose and baseline fasting insulin as covariates.
Time Frame: Baseline and Weeks 4, 8, 12, 16, 20, 26, 34, 42 and 52.
Population: as for outcome 13
Measure: Least Squares Mean (Standard Error); unit: μIU/mL
Arm/Group | Alogliptin 25 mg + Pioglitazone 30 mg + Metformin | Pioglitazone 45 mg + Metformin
Number analyzed (Participants) | 404 | 399
μIU/mL
  Week 4 (n=344, 328) | 0.53 (0.346) | -0.54 (0.355)
  Week 8 (n=382, 378) | 0.72 (0.393) | 0.05 (0.395)
  Week 12 (n=382, 378) | 1.21 (0.505) | 1.22 (0.507)
  Week 16 (n=383, 378) | 1.19 (0.414) | 0.56 (0.416)
  Week 20 (n=383, 378) | 1.60 (0.414) | 0.38 (0.417)
  Week 26 (n=383, 378) | 1.94 (0.479) | 0.88 (0.482)
  Week 34 (n=383, 378) | 1.41 (0.430) | 0.83 (0.433)
  Week 42 (n=383, 378) | 1.79 (0.441) | 1.10 (0.443)
  Week 52 (n=383, 378) | 1.91 (0.470) | 1.18 (0.473)
Statistical Analysis 1: Comparison: Alogliptin 25 mg + Pioglitazone 30 mg + Metformin vs Pioglitazone 45 mg + Metformin; Comparison of change from Baseline at Week 52; Test type: Superiority or Other; p = 0.276, ANCOVA — Statistical test and resulting P-value are 2-sided and was evaluated at the 0.05 significance level; ANCOVA model with treatment, study schedule and geographic region as class variables, and baseline metformin dose and fasting insulin as covariates; LS Mean Difference = 0.73, 95% CI 2-sided [-0.58 to 2.04]

15. Secondary Outcome: Change From Baseline in Proinsulin/Insulin Ratio
Description: The ratio of proinsulin to insulin was calculated as proinsulin (pmol/L) / insulin (μIU/mL) at weeks 4, 8, 12, 16, 20, 26, 34, 42 and 52 relative to the Baseline value. Least squares means were from an ANCOVA model with treatment, study schedule and geographic region as class variables, and baseline metformin dose and baseline fasting proinsulin/insulin ratio as covariates.
Time Frame: Baseline and Weeks 4, 8, 12, 16, 20, 26, 34, 42 and 52.
Population: as for outcome 13
Measure: Least Squares Mean (Standard Error); unit: ratio
Arm/Group | Alogliptin 25 mg + Pioglitazone 30 mg + Metformin | Pioglitazone 45 mg + Metformin
Number analyzed (Participants) | 404 | 399
ratio
  Week 4 (n=341, 325) | -0.046 (0.0095) | -0.005 (0.0097)
  Week 8 (n=380, 375) | -0.049 (0.0148) | -0.001 (0.0149)
  Week 12 (n=380, 375) | -0.053 (0.0105) | 0.004 (0.0106)
  Week 16 (n=381, 375) | -0.044 (0.0100) | 0.002 (0.0101)
  Week 20 (n=381, 375) | -0.037 (0.0085) | -0.004 (0.0085)
  Week 26 (n=381, 375) | -0.036 (0.0081) | -0.015 (0.0081)
  Week 34 (n=381, 375) | -0.038 (0.0084) | -0.004 (0.0085)
  Week 42 (n=381, 375) | -0.047 (0.0083) | -0.010 (0.0083)
  Week 52 (n=381, 375) | -0.048 (0.0080) | -0.007 (0.0081)
Statistical Analysis 1: Comparison: Alogliptin 25 mg + Pioglitazone 30 mg + Metformin vs Pioglitazone 45 mg + Metformin; Comparison of change from Baseline at Week 52; Test type: Superiority or Other; p < 0.001, ANCOVA — Statistical test and resulting P-value are 2-sided and was evaluated at the 0.05 significance level; Treatment, study schedule and geographic region as class variables, and baseline metformin dose and baseline proinsulin/insulin ratio as covariates; LS Mean Difference = -0.041, 95% CI 2-sided [-0.063 to -0.018]

16. Secondary Outcome: Change From Baseline in C-peptide
Description: C-peptide is a byproduct created when the hormone insulin is produced and is measured by a blood test. Change from Baseline was assessed at Weeks 4, 8, 12, 16, 20, 26, 34, 42 and 52. Least squares means are from an ANCOVA model with treatment, study schedule and geographic region as class variables, and baseline metformin dose and baseline fasting C-peptide as covariates.
Time Frame: Baseline and Weeks 4, 8, 12, 16, 20, 26, 34, 42 and 52.
Population: as for outcome 13
Measure: Least Squares Mean (Standard Error); unit: ng/mL
Arm/Group | Alogliptin 25 mg + Pioglitazone 30 mg + Metformin | Pioglitazone 45 mg + Metformin
Number analyzed (Participants) | 404 | 399
ng/mL
  Week 4 (n=349, 333) | 0.110 (0.0350) | -0.033 (0.0358)
  Week 8 (n=393, 389) | 0.074 (0.0387) | -0.038 (0.0389)
  Week 12 (n=394, 390) | 0.070 (0.0459) | 0.030 (0.0462)
  Week 16 (n=395, 390) | 0.064 (0.0380) | 0.010 (0.0382)
  Week 20 (n=395, 390) | 0.104 (0.0384) | -0.001 (0.0386)
  Week 26 (n=395, 390) | 0.102 (0.0407) | -0.013 (0.0409)
  Week 34 (n=395, 390) | 0.118 (0.0403) | 0.003 (0.0406)
  Week 42 (n=395, 390) | 0.140 (0.0413) | 0.037 (0.0415)
  Week 52 (n=395, 390) | 0.182 (0.0430) | 0.108 (0.0433)
Statistical Analysis 1: Comparison: Alogliptin 25 mg + Pioglitazone 30 mg + Metformin vs Pioglitazone 45 mg + Metformin; Comparison of change from Baseline at Week 52; Test type: Superiority or Other; p = 0.230, ANCOVA — Statistical test and resulting P-value are 2-sided and was evaluated at the 0.05 significance level; Treatment, study schedule and geographic region as class variables, and baseline metformin dose and baseline fasting C-peptide as covariates; LS Mean Difference = 0.073, 95% CI 2-sided [-0.047 to 0.193]

17. Secondary Outcome: Change From Baseline in Calculated HOMA Insulin Resistance
Description: The Homeostasis Model Assessment of insulin resistance (HOMA IR) measures insulin resistance based on fasting glucose and insulin measurements:
  HOMA IR = fasting plasma insulin (µIU/mL) * fasting plasma glucose (mmol/L) / 22.5
  A higher number indicates a greater degree of insulin resistance. The change from Baseline in HOMA IR was assessed at Weeks 12, 26, 42 and 52. Least squares means are from an ANCOVA model with treatment, study schedule and geographic region as class variables, and baseline metformin dose and baseline HOMA insulin resistance as covariates.
Time Frame: Baseline and Weeks 12, 26, 42 and 52.
Population: as for outcome 13
Measure: Least Squares Mean (Standard Error); unit: insulin resistance
Arm/Group | Alogliptin 25 mg + Pioglitazone 30 mg + Metformin | Pioglitazone 45 mg + Metformin
Number analyzed (Participants) | 404 | 399
insulin resistance
  Week 12 (n=380, 378) | 0.007 (0.2339) | 0.350 (0.2345)
  Week 26 (n=381, 378) | 0.336 (0.2446) | 0.312 (0.2455)
  Week 42 (n=381, 378) | 0.200 (0.2103) | 0.431 (0.2111)
  Week 52 (n=381, 378) | 0.353 (0.2310) | 0.541 (0.2319)
Statistical Analysis 1: Comparison: Alogliptin 25 mg + Pioglitazone 30 mg + Metformin vs Pioglitazone 45 mg + Metformin; Comparison of change from Baseline at Week 52; Test type: Superiority or Other; p = 0.567, ANCOVA — Statistical test and resulting P-value are 2-sided and was evaluated at the 0.05 significance level; Treatment, study schedule and geographic region as class variables, and baseline metformin dose and baseline HOMA insulin resistance as covariates; LS Mean Difference = -0.188, 95% CI 2-sided [-0.830 to 0.455]

18. Secondary Outcome: Change From Baseline in Calculated HOMA Beta-cell Function
Description: The Homeostasis Model Assessment (HOMA) estimates steady state beta cell function (%B) as a percentage of a normal reference population.
  HOMA %B = 20 * insulin (µIU/mL) / fasting plasma glucose (mmol/L) - 3.5
  The change from Baseline in the homeostasis model assessment of beta cell function was assessed at Weeks 12, 26, 42 and 52. Least squares means are from an ANCOVA model with treatment, study schedule and geographic region as class variables, and baseline metformin dose and baseline HOMA beta cell function as covariates.
Time Frame: Baseline and Weeks 12, 26, 42 and 52.
Population: as for outcome 13
Measure: Least Squares Mean (Standard Error); unit: percentage beta cell function
Arm/Group | Alogliptin 25 mg + Pioglitazone 30 mg + Metformin | Pioglitazone 45 mg + Metformin
Number analyzed (Participants) | 404 | 399
percentage beta cell function
  Week 12 (n=380, 377) | 14.770 (3.6543) | 4.580 (3.6689)
  Week 26 (n=381, 377) | 30.012 (8.6151) | 3.242 (8.6608)
  Week 42 (n=381, 377) | 15.397 (2.7628) | 2.400 (2.7774)
  Week 52 (n=381, 377) | 15.020 (2.7396) | 2.057 (2.7541)
Statistical Analysis 1: Comparison: Alogliptin 25 mg + Pioglitazone 30 mg + Metformin vs Pioglitazone 45 mg + Metformin; Comparison of change from Baseline at Week 52; Test type: Superiority or Other; p < 0.001, ANCOVA — Statistical test and resulting P-value are 2-sided and was evaluated at the 0.05 significance level; Treatment, study schedule and geographic region as class variables, and baseline metformin dose and baseline HOMA beta cell function as covariates; LS Mean Difference = 12.963, 95% CI 2-sided [5.333 to 20.592]

19. Secondary Outcome: Change From Baseline in Body Weight
Description: Change from Baseline in body weight was assessed at Weeks 4, 8, 12, 26, 42 and 52. Least squares means are from an ANCOVA model with treatment, study schedule and geographic region as class variables, and baseline metformin dose and baseline body weight as covariates.
Time Frame: Baseline and Weeks 4, 8, 12, 26, 42 and 52.
Population: as for outcome 13
Measure: Least Squares Mean (Standard Error); unit: kg
Arm/Group | Alogliptin 25 mg + Pioglitazone 30 mg + Metformin | Pioglitazone 45 mg + Metformin
Number analyzed (Participants) | 404 | 399
kg
  Week 4 (n=354, 344) | 0.18 (0.094) | 0.32 (0.095)
  Week 8 (n=394, 394 | 0.31 (0.107) | 0.51 (0.107)
  Week 12 (n=395, 394) | 0.35 (0.124) | 0.64 (0.124)
  Week 26 (n=395, 394) | 0.73 (0.150) | 0.97 (0.150)
  Week 42 (n=395, 394) | 1.09 (0.179) | 1.52 (0.179)
  Week 52 (n=395, 394) | 1.10 (0.194) | 1.60 (0.194)
Statistical Analysis 1: Comparison: Alogliptin 25 mg + Pioglitazone 30 mg + Metformin vs Pioglitazone 45 mg + Metformin; Comparison of change from Baseline at Week 52; Test type: Superiority or Other; p = 0.071, ANCOVA — Statistical test and resulting P-value are 2-sided and was evaluated at the 0.05 significance level; Treatment, study schedule and geographic region as class variables, and baseline metformin dose and baseline body weight as covariates; LS Mean Difference = -0.50, 95% CI 2-sided [-1.03 to 0.04]

20. Secondary Outcome: Change From Baseline in Total Cholesterol
Description: Change from Baseline in total cholesterol was assessed at Weeks 4, 8, 12, 16, 20, 26, 34, 42 and 52. Least squares means are from an ANCOVA model with treatment, study schedule and geographic region as class variables, and baseline metformin dose and baseline total cholesterol as covariates.
Time Frame: Baseline and Weeks 4, 8, 12, 16, 20, 26, 34, 42 and 52.
Population: as for outcome 13
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Alogliptin 25 mg + Pioglitazone 30 mg + Metformin | Pioglitazone 45 mg + Metformin
Number analyzed (Participants) | 404 | 399
mg/dL
  Week 4 (n=397, 393) | -5.2 (1.28) | -1.9 (1.29)
  Week 8 (n=399, 395) | -4.0 (1.40) | 0.3 (1.40)
  Week 12 (n=399, 395) | -3.6 (1.44) | 1.1 (1.45)
  Week 16 (n=399, 395) | -4.3 (1.56) | -0.4 (1.57)
  Week 20 (n=399, 395) | -3.9 (1.55) | -0.5 (1.56)
  Week 26 (n=399, 395) | -2.1 (1.62) | 1.0 (1.63)
  Week 34 (n=399, 395) | -3.5 (1.61) | -0.7 (1.62)
  Week 42 (n=399, 395) | -3.8 (1.62) | 0.0 (1.62)
  Week 52 (n=399, 395) | -4.4 (1.58) | -0.1 (1.59)
Statistical Analysis 1: Comparison: Alogliptin 25 mg + Pioglitazone 30 mg + Metformin vs Pioglitazone 45 mg + Metformin; Comparison of change from Baseline at Week 52; Test type: Superiority or Other; p = 0.058, ANCOVA — Statistical test and resulting P-value are 2-sided and was evaluated at the 0.05 significance level; Treatment, study schedule and geographic region as class variables, and baseline metformin dose and baseline total cholesterol as covariates; LS Mean Difference = -4.2, 95% CI 2-sided [-8.6 to 0.1]

21. Secondary Outcome: Change From Baseline in High-Density Lipoprotein Cholesterol
Description: Change from Baseline in high-density lipoprotein cholesterol (HDL-C) was assessed at Weeks 4, 8, 12, 16, 20, 26, 34, 42 and 52. Least squares means are from an ANCOVA model with treatment, study schedule and geographic region as class variables, and baseline metformin dose and baseline HDL cholesterol as covariates.
Time Frame: Baseline and Weeks 4, 8, 12, 16, 20, 26, 34, 42 and 52.
Population: as for outcome 13
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Alogliptin 25 mg + Pioglitazone 30 mg + Metformin | Pioglitazone 45 mg + Metformin
Number analyzed (Participants) | 404 | 399
mg/dL
  Week 4 (n=397, 392) | -0.7 (0.33) | 0.4 (0.34)
  Week 8 (n=399, 395) | -0.8 (0.35) | 0.6 (0.35)
  Week 12 (n=399, 395) | -0.2 (0.42) | 1.1 (0.42)
  Week 16 (n=399, 395) | -0.5 (0.37) | 0.9 (0.38)
  Week 20 (n=399, 395) | -0.2 (0.37) | 0.7 (0.37)
  Week 26 (n=399, 395) | 0.0 (0.37) | 0.6 (0.37)
  Week 34 (n=399, 395) | -0.6 (0.38) | 0.3 (0.38)
  Week 42 (n=399, 395) | -0.3 (0.38) | 0.6 (0.38)
  Week 52 (n=395, 395) | -0.3 (0.37) | 0.3 (0.37)
Statistical Analysis 1: Comparison: Alogliptin 25 mg + Pioglitazone 30 mg + Metformin vs Pioglitazone 45 mg + Metformin; Comparison of change from Baseline at Week 52; Test type: Superiority or Other; p = 0.228, ANCOVA — Statistical test and resulting P-value are 2-sided and was evaluated at the 0.05 significance level; Treatment, study schedule and geographic region as class variables, and baseline metformin dose and baseline HDL cholesterol as covariates; LS Mean Difference = -0.6, 95% CI 2-sided [-1.7 to 0.4]

22. Secondary Outcome: Change From Baseline in Low-Density Lipoprotein Cholesterol
Description: Change from Baseline in low-density lipoprotein cholesterol (LDL-C) was assessed at Weeks 4, 8, 12, 16, 20, 26, 34, 42 and 52. Least squares means are from an ANCOVA model with treatment, study schedule and geographic region as class variables, and baseline metformin dose and baseline LDL cholesterol as covariates.
Time Frame: Baseline and Weeks 4, 8, 12, 16, 20, 26, 34, 42 and 52.
Population: as for outcome 13
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Alogliptin 25 mg + Pioglitazone 30 mg + Metformin | Pioglitazone 45 mg + Metformin
Number analyzed (Participants) | 404 | 399
mg/dL
  Week 4 (n=388, 383) | -2.4 (1.11) | 0.0 (1.12)
  Week 8 (n=390, 386) | -0.6 (1.18) | 2.1 (1.19)
  Week 12 (n=390, 386) | -1.2 (1.21) | 1.4 (1.22)
  Week 16 (n=390, 386) | -1.7 (1.31) | -0.1 (1.32)
  Week 20 (n=390, 386) | -2.0 (1.24) | 0.1 (1.25)
  Week 26 (n=390, 386) | -0.6 (1.36) | 1.6 (1.37)
  Week 34 (n=390, 386) | -1.9 (1.33) | 1.2 (1.33)
  Week 42 (n=390, 386) | -1.6 (1.35) | 0.7 (1.36)
  Week 52 (n=390, 386) | -1.9 (1.32) | 1.0 (1.33)
Statistical Analysis 1: Comparison: Alogliptin 25 mg + Pioglitazone 30 mg + Metformin vs Pioglitazone 45 mg + Metformin; Comparison of change from Baseline at Week 52; Test type: Superiority or Other; p = 0.132, ANCOVA — Statistical test and resulting P-value are 2-sided and was evaluated at the 0.05 significance level; Treatment, study schedule and geographic region as class variables, and baseline metformin dose and baseline LDL cholesterol as covariates; LS Mean Difference = -2.8, 95% CI 2-sided [-6.5 to 0.9]

23. Secondary Outcome: Change From Baseline in Triglycerides
Description: Change from Baseline in triglycerides was assessed at Weeks 4, 8, 12, 16, 20, 26, 34, 42 and 52. Least squares means are from an ANCOVA model with treatment, study schedule and geographic region as class variables, and baseline metformin dose and baseline triglycerides as covariates.
Time Frame: Baseline and Weeks 4, 8, 12, 16, 20, 26, 34, 42 and 52.
Population: as for outcome 13
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Alogliptin 25 mg + Pioglitazone 30 mg + Metformin | Pioglitazone 45 mg + Metformin
Number analyzed (Participants) | 404 | 399
mg/dL
  Week 4 (n=397, 393) | -16.4 (2.98) | -12.2 (3.00)
  Week 8 (n=399, 395) | -17.9 (3.61) | -12.3 (3.63)
  Week 12 (n=399, 395) | -16.1 (3.69) | -4.5 (3.71)
  Week 16 (n=399, 395) | -16.3 (3.36) | -9.4 (3.38)
  Week 20 (n=399, 395) | -12.7 (3.68) | -8.5 (3.70)
  Week 26 (n=399, 395) | -11.9 (3.98) | -6.3 (4.00)
  Week 34 (n=399, 395) | -7.4 (3.98) | -8.1 (4.00)
  Week 42 (n=399, 395) | -14.6 (3.67) | -7.0 (3.69)
  Week 52 (n=399, 395) | -16.4 (3.47) | -7.8 (3.49)
Statistical Analysis 1: Comparison: Alogliptin 25 mg + Pioglitazone 30 mg + Metformin vs Pioglitazone 45 mg + Metformin; Comparison of change from Baseline at Week 52; Test type: Superiority or Other; p = 0.080, ANCOVA — Statistical test and resulting P-value are 2-sided and was evaluated at the 0.05 significance level; Treatment, study schedule and geographic region as class variables, and baseline metformin dose and baseline triglycerides as covariates; LS Mean Difference = -8.6, 95% CI 2-sided [-18.3 to 1.0]

24. Secondary Outcome: Change From Baseline in Free Fatty Acids
Description: Change from Baseline in free fatty acids was assessed at Weeks 12, 26, 42 and 52. Least squares means are from an ANCOVA model with treatment, study schedule and geographic region as class variables, and baseline metformin dose and baseline free fatty acids as covariates.
Time Frame: Baseline and Weeks 12, 26, 42, and 52.
Population: as for outcome 13
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Alogliptin 25 mg + Pioglitazone 30 mg + Metformin | Pioglitazone 45 mg + Metformin
Number analyzed (Participants) | 404 | 399
mmol/L
  Week 12 (n=355, 360) | -0.0526 (0.01037) | -0.0332 (0.01031)
  Week 26 (n=366, 368) | -0.0364 (0.01231) | -0.0162 (0.01228)
  Week 42 (n=367, 368) | -0.0243 (0.01083) | -0.0222 (0.01081)
  Week 52 (n=367, 368) | -0.0294 (0.01173) | 0.0019 (0.01171)
Statistical Analysis 1: Comparison: Alogliptin 25 mg + Pioglitazone 30 mg + Metformin vs Pioglitazone 45 mg + Metformin; Comparison of change from Baseline at Week 52; Test type: Superiority or Other; p = 0.059, ANCOVA — Statistical test and resulting P-value are 2-sided and was evaluated at the 0.05 significance level; Treatment, study schedule and geographic region as class variables, and baseline metformin dose and baseline free fatty acid as covariates; LS Mean Difference = -0.0314, 95% CI 2-sided [-0.0640 to 0.0012]

25. Secondary Outcome: Change From Baseline in Apolipoprotein A1
Description: Change from Baseline in Apolipoprotein A1 was assessed at Weeks 12, 26, 42 and 52. Least squares means are from an ANCOVA model with treatment, study schedule and geographic region as class variables, and baseline metformin dose and baseline apolipoprotein A1 as covariates.
Time Frame: Baseline and Weeks 12, 26, 42 and 52.
Population: as for outcome 13
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Alogliptin 25 mg + Pioglitazone 30 mg + Metformin | Pioglitazone 45 mg + Metformin
Number analyzed (Participants) | 404 | 399
mg/dL
  Week 12 (n=348, 355) | 0.5 (0.99) | 0.0 (0.98)
  Week 26 (n=359, 363) | 0.1 (0.95) | -0.9 (0.95)
  Week 42 (n=360, 363) | -2.1 (0.95) | -2.2 (0.95)
  Week 52 (n=360, 363) | -4.5 (0.99) | -4.4 (0.98)
Statistical Analysis 1: Comparison: Alogliptin 25 mg + Pioglitazone 30 mg + Metformin vs Pioglitazone 45 mg + Metformin; Comparison of change from Baseline at Week 52; Test type: Superiority or Other; p = 0.934, ANCOVA — Statistical test and resulting P-value are 2-sided and was evaluated at the 0.05 significance level; Treatment, study schedule and geographic region as class variables, and baseline metformin dose and baseline apolipoprotein A1 as covariates; LS Mean Difference = -0.1, 95% CI 2-sided [-2.9 to 2.6]

26. Secondary Outcome: Change From Baseline in Apolipoprotein A2
Description: Change from Baseline in Apolipoprotein A2 was assessed at Weeks 12, 26, 42 and 52. Least squares means are from an ANCOVA model with treatment, study schedule and geographic region as class variables, and baseline metformin dose and baseline apolipoprotein A2 as covariates.
Time Frame: Baseline and Weeks 12, 26, 42 and 52.
Population: as for outcome 13
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Alogliptin 25 mg + Pioglitazone 30 mg + Metformin | Pioglitazone 45 mg + Metformin
Number analyzed (Participants) | 404 | 399
mg/dL
  Week 12 (n=348, 355) | -0.4 (0.22) | 0.6 (0.22)
  Week 26 (n=359, 363) | 0.4 (0.23) | 0.7 (0.22)
  Week 42 (n=360, 363) | 0.8 (0.25) | 1.1 (0.25)
  Week 52 (n=360, 363) | 0.3 (0.24) | 1.0 (0.24)
Statistical Analysis 1: Comparison: Alogliptin 25 mg + Pioglitazone 30 mg + Metformin vs Pioglitazone 45 mg + Metformin; Comparison of change from Baseline at Week 52; Test type: Superiority or Other; p = 0.070, ANCOVA — Statistical test and resulting P-value are 2-sided and was evaluated at the 0.05 significance level; Treatment, study schedule and geographic region as class variables, and baseline metformin dose and baseline apolipoprotein A2 as covariates; LS Mean Difference = -0.6, 95% CI 2-sided [-1.3 to 0.1]

27. Secondary Outcome: Change From Baseline in Apolipoprotein B
Description: Change from Baseline in Apolipoprotein B was assessed at Weeks 12, 26, 42 and 52. Least squares means are from an ANCOVA model with treatment, study schedule and geographic region as class variables, and baseline metformin dose and baseline apolipoprotein B as covariates.
Time Frame: Baseline and Weeks 12, 26, 42 and 52.
Population: Full analysis set where Baseline and at least 1 postbaseline value were available. Last observation carried forward (LOCF) imputation was utilized.
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Alogliptin 25 mg + Pioglitazone 30 mg + Metformin | Pioglitazone 45 mg + Metformin
Number analyzed (Participants) | 404 | 399
mg/dL
  Week 12 [N=348, 355] | -3.1 (1.02) | 0.1 (1.01)
  Week 26 [N=359, 363] | -0.6 (1.09) | 1.1 (1.08)
  Week 42 [N=360, 363] | -0.4 (1.15) | 1.8 (1.15)
  Week 52 [N=360, 363] | -1.2 (1.10) | 1.7 (1.10)
Statistical Analysis 1: Comparison: Alogliptin 25 mg + Pioglitazone 30 mg + Metformin vs Pioglitazone 45 mg + Metformin; Comparison of change from Baseline at Week 52; Test type: Superiority or Other; p = 0.064, ANCOVA — Statistical test and resulting P-value are 2-sided and was evaluated at the 0.05 significance level; Treatment, study schedule and geographic region as class variables, and baseline metformin dose and baseline apolipoprotein B as covariates; LS Mean Difference = -2.9, 95% CI 2-sided [-5.9 to 0.2]

28. Secondary Outcome: Change From Baseline in Apolipoprotein C-III
Description: Change from Baseline in Apolipoprotein C-III was assessed at Weeks 12, 26, 42 and 52. Least squares means are from an ANCOVA model with treatment, study schedule and geographic region as class variables, and baseline metformin dose and baseline apolipoprotein C-III as covariates.
Time Frame: Baseline and Weeks 12, 26, 42 and 52.
Population: as for outcome 27
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Alogliptin 25 mg + Pioglitazone 30 mg + Metformin | Pioglitazone 45 mg + Metformin
Number analyzed (Participants) | 404 | 399
mg/dL
  Week 12 (n=352, 361) | -0.6 (0.15) | 0.1 (0.15)
  Week 26 (n=365, 369) | -0.1 (0.17) | 0.2 (0.17)
  Week 42 (n=366, 369) | -0.3 (0.17) | 0.2 (0.17)
  Week 52 (n=366, 369) | -0.5 (0.16) | 0.0 (0.16)
Statistical Analysis 1: Comparison: Alogliptin 25 mg + Pioglitazone 30 mg + Metformin vs Pioglitazone 45 mg + Metformin; Comparison of change from Baseline at Week 52; Test type: Superiority or Other; p = 0.022, ANCOVA — Statistical test and resulting P-value are 2-sided and was evaluated at the 0.05 significance level; Treatment, study schedule and geographic region as class variables, and baseline metformin dose and baseline apolipoprotein C-III as covariates; LS Mean Difference = -0.5, 95% CI 2-sided [-1.0 to -0.1]

29. Secondary Outcome: Change From Baseline in Plasminogen Activator Inhibitor-1
Description: Change from Baseline in plasminogen activator inhibitor-1 (PAI-1) was assessed at Weeks 12, 26, 42 and 52. Least squares means are from an ANCOVA model with treatment, study schedule and geographic region as class variables, and baseline metformin dose and baseline PAI-1 as covariates.
Time Frame: Baseline and Weeks 12, 26, 42 and 52.
Population: as for outcome 13
Measure: Least Squares Mean (Standard Error); unit: ng/ml
Arm/Group | Alogliptin 25 mg + Pioglitazone 30 mg + Metformin | Pioglitazone 45 mg + Metformin
Number analyzed (Participants) | 404 | 399
ng/ml
  Week 12 (n=322, 330) | -3.23 (1.483) | -3.59 (1.464)
  Week 26 (n=342, 343) | -2.83 (1.523) | -3.63 (1.520)
  Week 42 (n=346, 344) | -2.08 (1.429) | -4.89 (1.434)
  Week 52 (n=346, 344) | -2.92 (1.234) | -4.70 (1.237)
Statistical Analysis 1: Comparison: Alogliptin 25 mg + Pioglitazone 30 mg + Metformin vs Pioglitazone 45 mg + Metformin; Comparison of change from Baseline at Week 52; Test type: Superiority or Other; p = 0.308, ANCOVA — Statistical test and resulting P-value are 2-sided and was evaluated at the 0.05 significance level; Treatment, study schedule and geographic region as class variables, and baseline metformin dose and baseline PAI-1 as covariates; LS Mean Difference = 1.78, 95% CI 2-sided [-1.65 to 5.22]

30. Secondary Outcome: Change From Baseline in High-sensitivity C-Reactive Protein
Description: Change from Baseline in high-sensitivity C-Reactive Protein (hsCRP) was assessed at Weeks 12, 26, 42 and 52. Least squares means are from an ANCOVA model with treatment, study schedule and geographic region as class variables, and baseline metformin dose and baseline hsCRP as covariates.
Time Frame: Baseline and Weeks 12, 26, 42 and 52.
Population: as for outcome 13
Measure: Least Squares Mean (Standard Error); unit: mg/L
Arm/Group | Alogliptin 25 mg + Pioglitazone 30 mg + Metformin | Pioglitazone 45 mg + Metformin
Number analyzed (Participants) | 404 | 399
mg/L
  Week 12 (n=357, 366) | 0.2989 (0.53213) | 0.7049 (0.52569)
  Week 26 (n=366, 373) | -0.0632 (0.49229) | 0.9706 (0.48763)
  Week 42 (n=367, 373) | 0.7251 (0.48203) | 0.6443 (0.47813)
  Week 52 (n=367, 373) | 0.5875 (0.54194) | 1.4085 (0.53755)
Statistical Analysis 1: Comparison: Alogliptin 25 mg + Pioglitazone 30 mg + Metformin vs Pioglitazone 45 mg + Metformin; Comparison of change from Baseline at Week 52; Test type: Superiority or Other; p = 0.283, ANCOVA — Statistical test and resulting P-value are 2-sided and was evaluated at the 0.05 significance level; Treatment, study schedule and geographic region as class variables, and baseline metformin dose and baseline hsCRP as covariates; LS Mean Difference = -0.8209, 95% CI 2-sided [-2.3209 to 0.6790]

31. Secondary Outcome: Change From Baseline in Adiponectin
Description: Change from Baseline in adiponectin was assessed at Weeks 12, 26, 42 and 52. Least squares means are from an ANCOVA model with treatment, study schedule and geographic region as class variables, and baseline metformin dose and baseline adiponectin as covariates.
Time Frame: Baseline and Weeks 12, 26, 42 and 52.
Population: as for outcome 13
Measure: Least Squares Mean (Standard Error); unit: μg/mL
Arm/Group | Alogliptin 25 mg + Pioglitazone 30 mg + Metformin | Pioglitazone 45 mg + Metformin
Number analyzed (Participants) | 404 | 399
μg/mL
  Week 12 (n=355, 361) | 1.15 (0.453) | 2.97 (0.449)
  Week 26 (n=366, 371) | 1.17 (0.599) | 4.19 (0.595)
  Week 42 (n=367, 371) | -0.41 (0.529) | 3.04 (0.526)
  Week 52 (n=367, 371) | -0.70 (0.595) | 2.21 (0.591)
Statistical Analysis 1: Comparison: Alogliptin 25 mg + Pioglitazone 30 mg + Metformin vs Pioglitazone 45 mg + Metformin; Comparison of change from Baseline at Week 52; Test type: Superiority or Other; p < 0.001, ANCOVA — Statistical test and resulting P-value are 2-sided and was evaluated at the 0.05 significance level; Treatment, study schedule and geographic region as class variables, and baseline metformin dose and baseline adiponectin as covariates; LS Mean Difference = -2.92, 95% CI 2-sided [-4.57 to -1.27]

32. Secondary Outcome: Change From Baseline in Nuclear Magnetic Resonance Lipid Fractionation Total Triglycerides
Description: Nuclear Magnetic Resonance (NMR) lipid fractionation was used to assess the change from Baseline in total triglyceride levels at Weeks 12, 26, 42 and 52. Least squares means are from an ANCOVA model with treatment, study schedule and geographic region as class variables, and baseline metformin dose and baseline NMR triglycerides as covariates.
Time Frame: Baseline and Weeks 12, 26, 42 and 52.
Population: as for outcome 13
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Alogliptin 25 mg + Pioglitazone 30 mg + Metformin | Pioglitazone 45 mg + Metformin
Number analyzed (Participants) | 404 | 399
mg/dL
  Week 12 (n=357, 361) | -8.7 (3.24) | 0.2 (3.23)
  Week 26 (n=367, 368) | -1.7 (3.58) | 0.8 (3.58)
  Week 42 (n=367, 369) | -6.4 (3.60) | 0.7 (3.59)
  Week 52 (n=367, 369) | -6.9 (3.35) | -0.7 (3.34)
Statistical Analysis 1: Comparison: Alogliptin 25 mg + Pioglitazone 30 mg + Metformin vs Pioglitazone 45 mg + Metformin; Comparison of change from Baseline at Week 52; Test type: Superiority or Other; p = 0.197, ANCOVA — Statistical test and resulting P-value are 2-sided and was evaluated at the 0.05 significance level; LS Mean Difference = -6.1, 95% CI 2-sided [-15.4 to 3.2]

33. Secondary Outcome: Change From Baseline in Very Low Density Lipoprotein (VLDL) / Chylomicron Particles
Description: The change from Baseline in levels of total VLDL/chylomicron particles and large VLDL/chylomicron particles was assessed by NMR lipid fractionation at Weeks 12, 26, 42 and 52.
  Least squares means are from an ANCOVA model with treatment, study schedule and geographic region as class variables, and baseline metformin dose and baseline VLDL/chylomicron particles as covariates.
Time Frame: Baseline and Weeks 12, 26, 42 and 52.
Population: as for outcome 13
Measure: Least Squares Mean (Standard Error); unit: nmol/L
Arm/Group | Alogliptin 25 mg + Pioglitazone 30 mg + Metformin | Pioglitazone 45 mg + Metformin
Number analyzed (Participants) | 404 | 399
nmol/L
  Total Particles - Week 12 (n=357, 361) | -0.59 (1.814) | 2.39 (1.805)
  Total Particles - Week 26 (n=367, 368) | 1.27 (1.940) | 3.09 (1.937)
  Total Particles - Week 42 (n=367, 369) | -1.35 (1.916) | 1.64 (1.911)
  Total Particles - Week 52 (n=367, 369) | -1.20 (1.890) | 3.03 (1.885)
  Large Particles - Week 12 (n=357, 361) | -0.83 (0.247) | -0.27 (0.246)
  Large Particles - Week 26 (n=367, 368) | -0.39 (0.282) | -0.32 (0.281)
  Large Particles - Week 42 (n=367, 369) | -0.72 (0.277) | -0.38 (0.277)
  Large Particles - Week 52 (n=367, 369) | -0.66 (0.260) | -0.46 (0.260)

34. Secondary Outcome: Change From Baseline in VLDL / Chylomicron Triglycerides
Description: The change from Baseline in levels of VLDL/chylomicron triglycerides was assessed by NMR lipid fractionation at Weeks 12, 26, 42 and 52.
  Least squares means are from an ANCOVA model with treatment, study schedule and geographic region as class variables, and baseline metformin dose and baseline VLDL/chylomicron triglycerides as covariates.
Time Frame: Baseline and Weeks 12, 26, 42 and 52.
Population: as for outcome 13
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Alogliptin 25 mg + Pioglitazone 30 mg + Metformin | Pioglitazone 45 mg + Metformin
Number analyzed (Participants) | 404 | 399
mg/dL
  Week 12 (n=357, 361) | -7.6 (3.22) | -0.2 (3.20)
  Week 26 (n=367, 368) | -1.3 (3.54) | 0.2 (3.54)
  Week 42 (n=367, 369) | -5.4 (3.60) | 0.2 (3.59)
  Week 52 (n=367, 369) | -6.1 (3.30) | -1.5 (3.29)

35. Secondary Outcome: Change From Baseline in VLDL Particles
Description: The change from Baseline in levels of medium VLDL particles and small VLDL particles was assessed by NMR fractionation at Weeks 12, 26, 42 and 52. Least squares means are from an ANCOVA model with treatment, study schedule and geographic region as class variables, and baseline metformin dose and baseline VLDL particles as covariates.
Time Frame: Baseline and Weeks 12, 26, 42 and 52.
Population: as for outcome 13
Measure: Least Squares Mean (Standard Error); unit: nmol/L
Arm/Group | Alogliptin 25 mg + Pioglitazone 30 mg + Metformin | Pioglitazone 45 mg + Metformin
Number analyzed (Participants) | 404 | 399
nmol/L
  Medium Particles - Week 12 (n=357, 361) | -0.09 (1.152) | 1.74 (1.146)
  Medium Particles - Week 26 (n=367, 368) | 1.30 (1.208) | 2.23 (1.207)
  Medium Particles - Week 42 (n=367, 369) | 1.03 (1.307) | 2.43 (1.303)
  Medium Particles - Week 52 (n=367, 369) | 0.26 (1.166) | 2.12 (1.163)
  Small Particles - Week 12 (n=357, 361) | -0.04 (1.077) | 1.30 (1.072)
  Small Particles - Week 26 (n=367, 368) | 0.07 (1.121) | 1.47 (1.119)
  Small Particles - Week 42 (n=367, 369) | -1.86 (1.120) | -0.21 (1.117)
  Small Particles - Week 52 (n=367, 369) | -1.02 (1.192) | 1.58 (1.189)

36. Secondary Outcome: Change From Baseline in Mean VLDL Particle Size
Description: Change from Baseline in mean VLDL particle size was assessed by NMR lipid fractionation at Weeks 12, 26, 42 and 52. Least squares means are from an ANCOVA model with treatment, study schedule and geographic region as class variables, and baseline metformin dose and baseline mean VLDL particle size as covariates.
Time Frame: Baseline and Weeks 12, 26, 42 and 52.
Population: as for outcome 13
Measure: Least Squares Mean (Standard Error); unit: nm
Arm/Group | Alogliptin 25 mg + Pioglitazone 30 mg + Metformin | Pioglitazone 45 mg + Metformin
Number analyzed (Participants) | 404 | 399
nm
  Week 12 (n=355, 361) | -0.67 (0.369) | -0.79 (0.366)
  Week 26 (n=365, 368) | 0.11 (0.391) | -0.87 (0.389)
  Week 42 (n=365, 369) | 0.44 (0.445) | -0.79 (0.442)
  Week 52 (n=365, 369) | -0.12 (0.395) | -1.04 (0.393)

37. Secondary Outcome: Change From Baseline in Intermediate Density Lipoprotein (IDL) Particles
Description: The change from Baseline in levels of IDL particles was assessed by NMR lipid fractionation at Weeks 12, 26, 42 and 52. Least squares means are from an ANCOVA model with treatment, study schedule and geographic region as class variables, and baseline metformin dose and baseline IDL particles as covariates.
Time Frame: Baseline and Weeks 12, 26, 42 and 52.
Population: as for outcome 13
Measure: Least Squares Mean (Standard Error); unit: nmol/L
Arm/Group | Alogliptin 25 mg + Pioglitazone 30 mg + Metformin | Pioglitazone 45 mg + Metformin
Number analyzed (Participants) | 404 | 399
nmol/L
  Week 12 (n=357, 361) | -4.9 (2.24) | 3.2 (2.23)
  Week 26 (n=367, 368) | -4.1 (2.39) | 1.0 (2.39)
  Week 42 (n=367, 369) | -5.6 (2.26) | 2.0 (2.26)
  Week 52 (n=367, 369) | -4.5 (2.22) | 3.2 (2.21)

38. Secondary Outcome: Change From Baseline in Low Density Lipoprotein (LDL) Particles
Description: The change from Baseline in levels of total, large, medium-small, total small and very small LDL particles was assessed by NMR fractionation at Weeks 12, 26, 42 and 52. Least squares means are from an ANCOVA model with treatment, study schedule and geographic region as class variables, and baseline metformin dose and baseline LDL particles as covariates.
Time Frame: Baseline and Weeks 12, 26, 42 and 52.
Population: as for outcome 13
Measure: Least Squares Mean (Standard Error); unit: nmol/L
Arm/Group | Alogliptin 25 mg + Pioglitazone 30 mg + Metformin | Pioglitazone 45 mg + Metformin
Number analyzed (Participants) | 404 | 399
nmol/L
  Total Particles - Week 12 (n=357, 361) | -46.9 (14.88) | -22.3 (14.81)
  Total Particles - Week 26 (n=367, 368) | -14.0 (15.83) | -8.2 (15.81)
  Total Particles - Week 42 (n=367, 369) | -11.7 (16.86) | -10.7 (16.81)
  Total Particles - Week 52 (n=367, 369) | -13.0 (15.98) | -2.7 (15.94)
  Large Particles - Week 12 (n=357, 361) | -4.4 (9.29) | -5.0 (9.24)
  Large Particles - Week 26 (n=367, 368) | 1.1 (10.37) | 8.8 (10.36)
  Large Particles - Week 42 (n=367, 369) | -20.8 (9.68) | 0.0 (9.65)
  Large Particles - Week 52 (n=367, 369) | -19.2 (10.03) | -2.4 (10.00)
  Medium-small Particles - Week 12 (n=357, 361) | -7.0 (3.45) | -0.3 (3.43)
  Medium-small Particles - Week 26 (n=367, 368) | -0.7 (3.57) | -0.7 (3.57)
  Medium-small Particles - Week 42 (n=367, 369) | 4.1 (3.82) | 1.8 (3.81)
  Medium-small Particles - Week 52 (n=367, 369) | 2.4 (3.54) | 1.2 (3.53)
  Total Small Particles - Week 12 (n=357, 361) | -37.6 (16.93) | -20.8 (16.84)
  Total Small Particles - Week 26 (n=367, 368) | -10.9 (17.80) | -18.2 (17.77)
  Total Small Particles - Week 42 (n=367, 369) | 15.0 (18.63) | -13.0 (18.58)
  Total Small Particles - Week 52 (n=367, 369) | 10.9 (17.84) | -3.5 (17.79)
  Very Small Particles - Week 12 (n=357, 361) | -30.6 (13.84) | -20.6 (13.77)
  Very Small Particles - Week 26 (n=367, 368) | -10.1 (14.49) | -17.5 (14.47)
  Very Small Particles - Week 42 (n=367, 369) | 11.0 (15.13) | -14.9 (15.09)
  Very Small Particles - Week 52 (n=367, 369) | 8.6 (14.56) | -4.8 (14.52)

39. Secondary Outcome: Change From Baseline in Mean LDL Particle Size
Description: Change from Baseline in mean LDL particle size was assessed by NMR lipid fractionation at Weeks 12, 26, 42 and 52. Least squares means are from an ANCOVA model with treatment, study schedule and geographic region as class variables, and baseline metformin dose and baseline mean LDL particle size as covariates.
Time Frame: Baseline and Weeks 12, 26, 42 and 52.
Population: as for outcome 13
Measure: Least Squares Mean (Standard Error); unit: nm
Arm/Group | Alogliptin 25 mg + Pioglitazone 30 mg + Metformin | Pioglitazone 45 mg + Metformin
Number analyzed (Participants) | 404 | 399
nm
  Week 12 (n=357, 361) | 0.05 (0.031) | 0.06 (0.031)
  Week 26 (n=367, 368) | 0.03 (0.032) | 0.07 (0.032)
  Week 42 (n=367, 369) | -0.02 (0.032) | 0.05 (0.032)
  Week 52 (n=367, 369) | -0.04 (0.032) | 0.03 (0.032)

40. Secondary Outcome: Change From Baseline in High Density Lipoprotein (HDL) Particles
Description: The change from Baseline in levels of total, large, medium and small HDL particles was assessed by NMR fractionation at Weeks 12, 26, 42 and 52. Least squares means are from an ANCOVA model with treatment, study schedule and geographic region as class variables, and baseline metformin dose and baseline HDL particles as covariates.
Time Frame: Baseline and Weeks 12, 26, 42 and 52.
Population: as for outcome 13
Measure: Least Squares Mean (Standard Error); unit: μmol/L
Arm/Group | Alogliptin 25 mg + Pioglitazone 30 mg + Metformin | Pioglitazone 45 mg + Metformin
Number analyzed (Participants) | 404 | 399
μmol/L
  Total Particles - Week 12 (n=357, 361) | -0.18 (0.224) | -0.14 (0.223)
  Total Particles - Week 26 (n=367, 368) | 0.37 (0.228) | 0.03 (0.227)
  Total Particles - Week 42 (n=367, 369) | 0.09 (0.227) | -0.11 (0.227)
  Total Particles - Week 52 (n=367, 369) | 0.38 (0.227) | 0.02 (0.226)
  Large Particles - Week 12 (n=357, 361) | 0.08 (0.102) | 0.35 (0.101)
  Large Particles - Week 26 (n=367, 368) | 0.19 (0.103) | 0.53 (0.103)
  Large Particles - Week 42 (n=367, 369) | 0.06 (0.102) | 0.51 (0.101)
  Large Particles - Week 52 (n=367, 369) | 0.19 (0.105) | 0.57 (0.105)
  Medium Particles - Week 12 (n=357, 361) | 0.10 (0.165) | 0.43 (0.164)
  Medium Particles - Week 26 (n=367, 368) | 0.71 (0.178) | 0.90 (0.178)
  Medium Particles - Week 42 (n=367, 369) | 0.57 (0.172) | 0.70 (0.171)
  Medium Particles - Week 52 (n=367, 369) | 0.66 (0.180) | 0.96 (0.179)
  Small Particles - Week 12 (n=357, 361) | -0.38 (0.243) | -0.92 (0.242)
  Small Particles - Week 26 (n=367, 368) | -0.53 (0.250) | -1.39 (0.250)
  Small Particles - Week 42 (n=367, 369) | -0.54 (0.247) | -1.31 (0.246)
  Small Particles - Week 52 (n=367, 369) | -0.47 (0.251) | -1.49 (0.250)

41. Secondary Outcome: Change From Baseline in Mean HDL Particle Size
Description: Change from Baseline in mean HDL particle size was assessed by NMR lipid fractionation at Weeks 12, 26, 42 and 52. Least squares means are from an ANCOVA model with treatment, study schedule and geographic region as class variables, and baseline metformin dose and baseline mean HDL particle size as covariates.
Time Frame: Baseline and Weeks 12, 26, 42 and 52.
Population: as for outcome 13
Measure: Least Squares Mean (Standard Error); unit: nm
Arm/Group | Alogliptin 25 mg + Pioglitazone 30 mg + Metformin | Pioglitazone 45 mg + Metformin
Number analyzed (Participants) | 404 | 399
nm
  Week 12 (n=357, 361) | 0.04 (0.012) | 0.05 (0.012)
  Week 26 (n=367, 368) | 0.04 (0.012) | 0.07 (0.012)
  Week 42 (n=367, 369) | 0.02 (0.012) | 0.07 (0.012)
  Week 52 (n=367, 369) | 0.03 (0.012) | 0.08 (0.012)

ADVERSE EVENTS:
Time Frame: Collection of AEs began from time of informed consent until the end of the study (Week 54 or End-of-Treatment/Early Termination) and from spontaneous reporting up to 30 days after the final dose of study drug.
Description: At each study visit, the investigator assessed whether any events had occurred. Patients could report events at any other time during the study. All events, whether reported by the patient or observed by the investigator, were documented, whether or not the investigator concluded the event to be related to the drug treatment.
Arm/Group | Alogliptin 25 mg + Pioglitazone 30 mg + Metformin | Pioglitazone 45 mg + Metformin
Serious Adverse Events (participants affected / at risk) | 20/404 | 20/399
Other Adverse Events (participants affected / at risk) | 116/404 | 104/399
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Alogliptin 25 mg + Pioglitazone 30 mg + Metformin (N=404) | Pioglitazone 45 mg + Metformin (N=399)
Acute myocardial infarction (Cardiac disorders) | 0 | 2
Angina unstable (Cardiac disorders) | 1 | 1
Coronary artery disease (Cardiac disorders) | 1 | 1
Myocardial infarction (Cardiac disorders) | 1 | 0
Acute vestibular syndrome (Ear and labyrinth disorders) | 1 | 0
Cataract (Eye disorders) | 0 | 2
Ocular myasthenia (Eye disorders) | 0 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 2 | 0
Abdominal abscess (Infections and infestations) | 0 | 1
Appendicitis (Infections and infestations) | 1 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 1
Hepatitis B (Infections and infestations) | 0 | 1
Lobar pneumonia (Infections and infestations) | 1 | 0
Osteomyelitis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1
Pneumonia primary atypical (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 2
Frostbite (Injury, poisoning and procedural complications) | 1 | 0
Injury (Injury, poisoning and procedural complications) | 1 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0
Wound dehiscence (Injury, poisoning and procedural complications) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Rectosigmoid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 1 | 0
Ischaemic stroke (Nervous system disorders) | 0 | 1
Migraine (Nervous system disorders) | 1 | 0
Mania (Psychiatric disorders) | 1 | 0
Calculus urinary (Renal and urinary disorders) | 0 | 1
Renal colic (Renal and urinary disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypotension (Vascular disorders) | 0 | 2
Arteriosclerosis obliterans (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 0 | 1
Peripheral vascular disorder (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Alogliptin 25 mg + Pioglitazone 30 mg + Metformin (N=404) | Pioglitazone 45 mg + Metformin (N=399)
Nasopharyngitis (Infections and infestations) | 28 | 21
Hypertension (Vascular disorders) | 24 | 21
Upper respiratory tract infection (Infections and infestations) | 29 | 16
Influenza (Infections and infestations) | 18 | 23
Diarrhoea (Gastrointestinal disorders) | 11 | 24
Urinary tract infection (Infections and infestations) | 22 | 13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.